CLINICAL TRIAL: NCT00807196
Title: Phase I-II Non-Randomized Study of Yttrium 90 Ibritumomab Tiuxetan (Zevalin) With Non Myeloablative Allogeneic Stem Cell Transplantation in Patients With Relapsed, Refractory, or Transformed Indolent Non Hodgkin Lymphoma
Brief Title: Zevalin With Non Myeloablative Allogeneic Stem Cell Transplantation in Patients With Non Hodgkin Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Carole Deschambault/executive director, Hopital Maisonneuve-Rosemont
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZEV0701
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Non-Hodgkins Lymphoma
Keywords: Allogeneic Stem Cell Transplantation; Zevalin; Non-Hodgkins Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; ibritumomab tiuxetan; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- T (Experimental)
  Interventions: Drug: Rituximab; Drug: 90Y ibritumomab tiuxetan (Zevalin); Drug: Cyclophosphamide; Drug: Fludarabine; Other: Non myeloablative allogeneic stem cell transplantation

INTERVENTIONS:
Drug: Rituximab — 250mg/m2 day -21 and day -14 of preparative regimen
Drug: 90Y ibritumomab tiuxetan (Zevalin) — 0.4 mCi/kg IV on day -14 of preparative regimen
Drug: Cyclophosphamide — 300mg/m2 IV daily for 5 days day -8 to day -4 of preparative regimen
Drug: Fludarabine — 30mg/m2 IV daily for 5 days day -8 to day -4 of preparative regimen
Other: Non myeloablative allogeneic stem cell transplantation — Blood stem cell infusion on day 0

SUMMARY:
The purpose of this study is to investigate the ability to combine a radioactive medication directly targeted against lymphoma cells with the immune effects of an allogeneic blood stem cell transplant.

DETAILED DESCRIPTION:
Despite initial high response rates of low grade Non Hodgkin lymphoma, progressive or refractory disease currently remains incurable. Being a radiosensitive tumor, we hypothesize that combining different modalities of treatment including targeted radioimmunotherapy (RIT), and a graft versus lymphoma effect related to an allogeneic non myeloablative stem cell transplant may increase response and survival rates in a safe manner in patients with persistent disease following initial treatment. In this study patients who are not eligible for a standard stem cell transplant approach because of relapsed or refractory disease and who have a related sibling donor are treated with RIT followed by an allogeneic non myeloablative blood stem cell transplant

ELIGIBILITY:
Inclusion Criteria:

Patients must have/be

1. Age 18 to 65 years. Patients between age 66 and 69 may be enrolled if judged to be in excellent physical condition as per treating physician and study investigator and based on institutional practice.
2. Diagnosis of Non-Hodgkin lymphoma, follicular, marginal zone, small lymphocytic lymphoma, mantle cell lymphoma or transformed from an indolent NHL to aggressive histology disease lymphoma as defined by the World Health Organization.
3. Disease relapsed after, refractory or failing to achieve a PR after two or more cycles of intensive salvage chemotherapy (R-ESHAP or other) or disease relapsed after autologous stem cell transplantation. Poor partial response is defined as less than 50% reduction of tumor size. Salvage chemotherapy has to be administered after either 1st, 2nd or 3rd relapse
4. Disease expressing the CD 20 antigen
5. ECOG performance status 0-2
6. Judged to be able to tolerate NST and Zevalin treatment based on institutional criteria.
7. Signed written informed consent
8. At least one fully HLA matched sibling without evident contraindications to the donation procedures and willing to sign consent for donation

Exclusion Criteria:

Patients must not have/be

1. Abnormal renal function (creatinine > 1.5 x upper limit of normal (ULN)
2. Abnormal hepatic function (bilirubin > 2 x ULN, ALT/AST>2x ULN)
3. Cardiac ejection fraction <40% and/or other significant cardiac compromise
4. Severe defects in pulmonary function tests or receiving continuous oxygen
5. Severe concurrent illness, such as symptomatic congestive heart failure, severe arrhythmias, uncontrolled hypertension, diabetes, severe neurologic or psychiatric disorder or known HIV positive
6. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1) that may impact on patients life expectancy or any cancer curatively treated < 3 years prior to study entry.
7. History of prior allogeneic bone marrow transplant
8. Evidence of active hepatitis B or C infection or positivity for hepatitis-B surface antigen
9. Known type 1 hypersensitivity or anaphylactic proteins to any component of the Zevalin therapy or a history or presence of human anti-mouse antibodies (HAMA)
10. A female patient who is pregnant or breast feeding and an adult of reproductive potential who is not employing an effective method of birth control during the study.
11. CNS lymphoma
12. Ongoing confirmed or suspected significant infection
13. Prior treatment with radioimmunotherapy
14. Other condition preventing participation in standard NST
15. No fully matched sibling donor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Engraftment, chimerism, transplant related toxicity, acute and chronic GVHD | one year

SECONDARY OUTCOMES:
Overall response rate, overall and disease free survival | 360 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kiss, MD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Hopital Maisonneuve-Rosemont, Montreal, Quebec, Canada